CLINICAL TRIAL: NCT03485703
Title: Randomized Clinical Trial: Use of Azithromycin to Prevent Lung Damage in Preterm Newborns Under Mechanical Ventilation
Brief Title: Azithromycin in the Prevention of Lung Injury in Premature Newborn
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110639
Record Dates: First submitted 2018-03-25; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: for a period of 5 days, a group of infants will receive azithromycin EV at a dose of 10 mg / kg / day and another group will receive placebo (SF 0.9%) in the same volume, every 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- azithromycin group (Experimental): A control group composed of 40 newborns receiving azithromycin
  Interventions: Drug: Azithromycin
- placebo group (Placebo Comparator): comparative group composed of 40 newborns who would receive saline 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — the newborn group will receive intravenous azithromycin 10 mg / kg / day once daily for 5 days
  Other Names: group A
  Arms: azithromycin group
Drug: Placebo — the group of newborns will receive 0.9% saline once daily for 5 days
  Other Names: group B
  Arms: placebo group

SUMMARY:
The introduction of invasive mechanical ventilation in the treatment of preterm infants works as an adjuvant in the treatment of acute respiratory failure, which has resulted in significantly significant survival rates. In recent years there has been an increase in the number of evidence that mechanical factors can cause lung injury through inflammatory cells and soluble mediators.

The alveolar and airway epithelium is an important source of cytokine release. Cytokines are very low molecular weight proteins or glycoproteins with hormone-like actions. They contribute to the pathogenesis of various diseases through the ability to induce other inflammatory mediators Mechanical ventilation strategies can increase pulmonary and systemic cytokines and lead to dysfunction of multiple organs and systems.

Azithromycin has a potent anti-inflammatory and immunomodulatory effect It suppresses the production of proinflammatory cytokines (IL-6, IL-1, and TNF-α), has effective antimicrobial properties against Ureaplasma and, best of all, few side effects The hypothesis of this study is that azithromycin would reduce pulmonary inflammation induced by mechanical ventilation in premature infants, conferring a protective character.Randomized clinical trial: use of azithromycin in preventing pulmonary damage newborn preterm undergoing mechanical ventilation

DETAILED DESCRIPTION:
The nature of lung injury induced by mechanical ventilation is clearly established, including the release of immunoinflammatory mediators. However, safe drug therapy that decreases its severity is not available. Azithromycin is a macrolide antibiotic with potent anti-inflammatory effects, but has been poorly studied in preterm infants except for very few studies in extreme preterms for the prevention of bronchopulmonary dysplasia.

The aim of this study was to evaluate the effect of azithromycin on the prevention of cytokine-mediated MV-induced injury in cytokine plasma levels (IL-1β, IL-2, IL-6, IL-8, IL-10 and TNF- α) in preterm newborns, submitted to mechanical ventilation in the first 72 hours of life.

It is a double-blind placebo controlled clinical trial. When the use of azithromycin was considered, after signing the informed consent, a randomization was performed by the intravenous mixtures center of Hospital de clinicas de porto alegre where a group of newborns will receive azithromycin EV at the dose of 10mg / kg / day and another group will receive placebo (SF 0.9%) in the same volume, a blood aliquot of 300μL will be collected in all ETDA for cytokine analysis and PCR for Ureaplasma. After 5 days of starting azithromycin or placebo, a new sample will be collected for cytokines along with blood collection from the patient's routine. There will be no blood collection exclusively for the study.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants of less than 37 weeks of gestational age who have undergone mechanical ventilation within the first 72 hours of life

Exclusion Criteria:

* Major congenital malformations or chromosomal syndromes Mothers carrying the HIV virus.

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-08-28 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-04-13 (Actual)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia | 28 days
  neonate that needs to use oxygen in concentrations above 21% for a period greater than or equal to 28 days

SECONDARY OUTCOMES:
TNF | 5 days
  decreasing in plasma levels after treatment with azitromicina
IL-10 | 5 days
  increasing in plasma levels after treatment with azitromicina
IL-6 | 5 days
  increasing in plasma levels after treatment with azitromicina
IL-8 | 5 days
  increasing in plasma levels after treatment with azitromicina
IL1b | 5 days
  increasing in plasma levels after treatment with azitromicina
IL2 | 5days
  increasing in plasma levels after treatment with azitromicina

CONTACTS AND LOCATIONS:
Overall Officials: Rita de Cassia Silveira, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nunes CR, Procianoy RS, Corso AL, Silveira RC. Use of Azithromycin for the Prevention of Lung Injury in Mechanically Ventilated Preterm Neonates: A Randomized Controlled Trial. Neonatology. 2020;117(4):522-528. doi: 10.1159/000509462. Epub 2020 Sep 7. PMID 32894857